CLINICAL TRIAL: NCT01956981
Title: Comparison Between Magnesium Sulfate and Dexmedetomidine in Controlled Hypotension During Functional Endoscopic Sinus Surgery: A Double-blind, Randomized Clinical Trial
Brief Title: Controlled Hypotension During Functional Endoscopic Sinus Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Adnan Bayram, Assisstant Professor, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2011-221
Record Dates: First submitted 2013-09-28; First posted 2013-10-08 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: Hemorrhage
Keywords: controlled hypotension, dexmedetomidine, magnesium sulfate.
MeSH Terms: conditions — Hemorrhage | interventions — Magnesium Sulfate; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Magnesium (Placebo Comparator): 40 mg kg-1 IV magnesium sulfate (OSEL ilaç San. Ve Tic. A.Ş., Beykoz, Istanbul, Turkey) in 100 ml saline solution was applied to patients in Group M as a loading dose 10 minutes before the induction and continued during the surgery at the dose of 10-15 mg kg-1hour-1.
  Interventions: Drug: Magnesium Sulfate
- Dexmedetomidine (Active Comparator): 1 µg kg-1 IV dexmedetomidine (Precedex Abbott Labs, North Chicago, IL) in 100 ml saline solution was applied to patients in group D 10 minutes before the surgery and continued during the surgery at the dose of 0.5-1 µg kg-1.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Magnesium Sulfate — 40 mg kg-1 IV magnesium sulfate (OSEL ilaç San. Ve Tic. A.Ş., Beykoz, Istanbul, Turkey) in 100 ml saline solution was applied to patients in Group M as a loading dose 10 minutes before the induction and continued during the surgery at the dose of 10-15 mg kg-1hour-1.
  Arms: Magnesium
Drug: Dexmedetomidine — 1 µg kg-1 IV dexmedetomidine (Precedex Abbott Labs, North Chicago, IL) in 100 ml saline solution was applied to patients in group D 10 minutes before the surgery and continued during the surgery at the dose of 0.5-1 µg kg-1.
  Other Names: Precedex
  Arms: Dexmedetomidine

SUMMARY:
It is very important to decrease the bleeding during functional endoscopic sinus surgery (FESS) in order to increase the visibility of the surgical site. Our primary goal was to investigate the effects of magnesium sulfate and dexmedetomidine used for controlled hypotension on visibility of surgical site.

DETAILED DESCRIPTION:
Background: It is very important to decrease the bleeding during functional endoscopic sinus surgery (FESS) in order to increase the visibility of the surgical site. Our primary goal was to investigate the effects of magnesium sulfate and dexmedetomidine used for controlled hypotension on visibility of surgical site.

Methods: Sixty patients aged between 18-65 years were enrolled. Patients were divided into two groups. In the magnesium sulfate group (Group M) patients were administered 40 kg-1 magnesium sulfate in 100 ml saline solution in 10 minutes as IV loading dose 10 minutes before the induction and 10-15 mgkg-1hour-1 infusion during the surgery. In the dexmedetomidine group (Group D) patients were administered 1 µgkg-1 dexmedetomidine in 100 ml saline solution as loading dose 10 minutes before the surgery and 0.5-1 µgkg-1hour-1 dexmedetomidine during the surgery. Deliberate hypotension was defined as a mean arterial pressure (MAP) being 60-70 mmHg.

ELIGIBILITY:
Inclusion Criteria:

18 and 65 years scheduled for functional endoscopic sinus surgery

Exclusion Criteria:

* Patients with kidney, liver, hematological and neuromuscular diseases, diabetic neuropathy, any known allergy history to studied agents.
* weight exceeding the ideal body weight more than 30%,
* Being treated with calcium channel blockers, non-steroidal anti-inflammatory drugs, agents affecting neuromuscular blockage,and agents contraindicated for controlled hypotension

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-01; Primary Completion 2013-03 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
visibility scale of the surgical site | every 5 minutes during surgery up to 60 minutes
  Surgical site was rated according to 6 point scale at every 5 minutes by the same surgeon in terms of bleeding and dryness during surgery

SECONDARY OUTCOMES:
Blood Pressure | up to 24 hours
  After the patients were taken to the operating room, mean arterial pressure (MAP)was monitored and data was measured at every 5 minutes. Hemodynamic data were recorded at the initial phase, after the induction, 5, 10, 15, 30 and 45 minutes after the intubating, 1 and 5 minutes after the extubating.

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Bayram, Asst. Prof., Study Chair — TC Erciyes University